CLINICAL TRIAL: NCT01890824
Title: The Effect of Chemotherapy on Fat Metabolism and Digestion and Function in Breast Cancer Patients.
Brief Title: Fat Metabolism Following Chemotherapy in Breast Cancer
Status: Terminated | Type: Observational
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Ph.D., Texas A&M University
Other Study IDs: 2013-0297F
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Fat metabolism; Fat digestion; physical activity; muscle function
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, adipose tissue, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breast Cancer Patients: Breast cancer patients to be studied before and after chemotherapy
- Healthy Female Controls: Healthy female controls will be compared to breast cancer patients before and after chemotherapy and to healthy male controls
- Healthy Male Controls: Healthy male controls will be compared to healthy female controls to determine gender differences

SUMMARY:
Following chemotherapy, breast cancer patients primarily gain fat mass and lose muscle mass. Both depletion of muscle and an increase of fat mass in breast cancer patients are related to short survival, and decreased skeletal muscle mass and function may result in fatigue and inactivity, which contributes to fat mass changes and can be responsible for chemo-toxicity and increased mortality. The purpose of this study is to provide detailed insight in chemotherapy related changes in lipid metabolism and gut digestion and absorption of fat in breast cancer patients compared to matched healthy controls. This will provide required information that is necessary to implement new strategies to develop optimal nutritional regimen in breast cancer patients. The hypothesis is that chemotherapy in breast cancer is related to altered gut function and absorption and to increases in fat synthesis that lead to fat accumulation. In addition, we will examine the effect of cancer, chemotherapy, and gender by comparing fat digestion/absorption and fat metabolism of the breast cancer before and after chemotherapy, to aged matched healthy female and male controls.

DETAILED DESCRIPTION:
This research study involves 5 visits for the breast cancer subjects and 3 visits for the healthy controls. The first visit includes the informed consent and a screening and the second and third visit for the study days before chemotherapy and the fourth and fifth visit for the study days after chemotherapy. For the first test day, 2 hours of the subjects time will be for urine and blood sample collection, and to ingest the deuterated water. Subjects are allowed to go home after and eat normally. On the second study day, subjects will arrive early that morning and a DXA scan will be performed first. For the duration of the study, subjects have to lie in the bed (except for bathroom privileges). They can watch tv or bring and use a book/tablet. The research nurse or study staff will be present in the human subject area to assist the subject if necessary. Subjects are not allowed to eat or drink during the second test day, except for the test drink (meal) and water. One IV catheter will be placed in a vein of the arm/hand for blood draws. The hand will be placed in a hot box during blood collection. Another IV catheter will be placed in the contra-lateral forearm for a primed and continuous infusion of 2H5-glycerol. Over the two day time period, a total of 100-120 ml of blood will be obtained over approximately 19 samples. Stable isotopes will be ingested on the first test day, added to the test drinks on the second test day after the second hour, and infused on the second day. On the second test day, subjects will fill out questionnaires and perform muscle function tests. After completion of the study, we will provide the subject with a meal.

ELIGIBILITY:
Inclusion criteria cancer subjects:

* Diagnosed with breast cancer
* Scheduled for chemotherapy
* Ability to sign informed consent
* Age 30 years and older
* Ability to lie in supine position for 7 hours

Inclusion criteria healthy subjects:

* Healthy male & female according to the investigator's or appointed staff's judgment
* Age 30 years or older
* No diagnosis of cancer

Exclusion Criteria:

* Presence of fever within the last 3 days
* Untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Use of nutritional supplements within 5 days of first test day
* Any other condition according to the PI or nurse that would interfere with the study or safety of the patient
* Failure to give informed consent
* Possible) pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with breast cancer will be recruited when visiting a medical or cancer clinic in and outside the surrounding area of College Station. Cancer patients and healthy subjects will also be recruited by responding to distributed flyers in the community in the College Station area; for example in hospital/clinic waiting areas, clinic rooms and bulletin boards at Scott & White and the CSMC or any other hospital. Other general recruitment material in relation to the nutrition research that the research group performs at Texas A&M can be placed on bulletin boards at Scott & White and the CSMC.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Hepatic triglyceride synthesis | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in hepatic triglyceride synthesis before and after a meal
Hepatic de novo lipogenesis | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in hepatic de novo lipogenesis before and after a meal

SECONDARY OUTCOMES:
Adipose tissue triglyceride synthesis | pre and 4 hours post meal
  changes in adipose tissue triglyceride synthesis before and after a meal
Adipose tissue de novo lipogenesis | pre and 4 hours post meal
  changes in adipose tissue de novo lipogenesis before and after a meal
Adipose tissue lipolysis - glycerol rate of appearance | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  changes in adipose tissue lipolysis before and after a meal. plasma enrichment of glycerol.
Fat digestion and absorption | Pre meal ingestion and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210, 240, 270, and 300 min post meal ingestion
  defining fat digestion and absorption after a meal. Enrichment in palmitic acid and tripalmitin fatty acids in plasma
Skeletal muscle strength and endurance | 1 day
  Difference in leg strength and fatigue
Insulin response to feeding | pre and up to 5 hours post meal
  acute changes from postabsorptive state to postprandial state
Body composition | 1 day
  body composition will be determined by dual-energy X-ray absorptiometry and by deuterated water dilution technique. Plasma deuterium enrichments will be determined.
Physical activity questionnaire | 1 day
  Outcome of physical activity assessment in breast cancer patients and healthy controls in relation to the fat metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Ph.D., Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States